CLINICAL TRIAL: NCT00671996
Title: A Local Feasibility Study on Mangafodipir as an Adjunct to FOLFOX6 Chemotherapy in Patients Operated Upon Colon Cancer Stage Dukes' C
Brief Title: Mangafodipir as an Adjunct to FOLFOX6 Chemotherapy in Colon Cancer Stage Dukes' C
Acronym: MANFOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Egetis Therapeutics (Industry)
Responsible Party: Jan Olof G. Karlsson, PledPharma AB, Grev Turegatan 7, SE-11446 Stockholm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PP 01-07
Record Dates: First submitted 2008-05-04; First posted 2008-05-06 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-05

CONDITIONS: Chemotherapy; Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — N,N'-bis(pyridoxal-5-phosphate)ethylenediamine-N,N'-diacetic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Mangafodipir treatment
  Interventions: Drug: Mangafodipir
- B (Placebo Comparator)
  Interventions: Drug: Placebo treatment (0.9% NaCl)

INTERVENTIONS:
Drug: Mangafodipir — Treatment will be undertaken with a ready-to-use investigative drug formulation identical to what is in diagnostic use as a contrast medium for MRI.
  Formulation content: MnDPDP 10 mmol/ml
  Administered dose per cycle: 2 μmol/kg b.w. Administration form: Ready-to-use formulation (solution). Mangafodipir or placebo (0.2 ml/kg b.w.) will be administered as an i.v. infusion over 5 min about 30 min prior to start of chemotherapy.
  Other Names: Teslascan; ACT code V08CAE05
  Arms: A
Drug: Placebo treatment (0.9% NaCl) — Intravenous infusion, 2 micromol/kg, pretreatment 30 minutes before the start of FOLFOX treatment (during the first three FOLFOX treatments)
  Arms: B

SUMMARY:
The present feasibility study is designed to find out whether pre-treatment with the compound mangafodipir lowers the frequency and severity of side effects during adjuvant chemotherapy according to the FOLFOX6 regimen in patients operated upon colon cancer in stage Dukes' C.

DETAILED DESCRIPTION:
Mangafodipir, manganese (Mn) dipyridoxyl diphosphate, is a catalytic antioxidant and iron chelator recently (2006) suggested for cancer treatment in an Editorial in Journal of the National Cancer Institute. Preclinical research has shown that mangafodipir protects normal tissues without loss of anti-tumour activity during chemotherapy. Other advantages are that mangafodipir is already approved for use in patients as a contrast agent for magnetic resonance imaging (MRI) of liver, and that the experience for more than a decade reveals high safety with mainly minor and tolerable side-effects.

The present study will include 14 patients who will be followed throughout 3 treatment cycles. Each cycle will be preceded by infusion of mangafodipir or placebo in two groups, each consisting of 7 patients. The primary endpoints will be the most frequent manifestation of FOLFOX6, namely neutropenia and neurosensory toxicity. The secondary endpoints will be the frequency and severity of other FOLFOX6-related adverse events and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven colon cancer stage Dukes' C.
2. Patient over 18 years.
3. WHO performance status <1.
4. Adequate haematological function (Hb ≥ 100 g/L, ANC ≥ 2.0 x 109/L, platelets ≥ 150 x 109/L)
5. Adequate renal and hepatic functions: serum creatinine and total bilirubin ≤ 1.25 times upper normal limits (ASAT and ALAT ≤ 3 times upper normal limits)
6. Clinical evaluation, haematology and biochemistry performed within 1 week prior to the start of chemotherapy
7. Use of adequate contraception (males with reproductive potential)
8. Written informed consent given

Exclusion Criteria:

1. Other tumour types than colon adenocarcinomas
2. Current severe neutropenia, leucopenia or thrombocytopenia
3. Severely reduced liver or renal function
4. Unresolved bowel obstruction or sub-obstruction, uncontrolled Crohn's disease or ulcerative colitis
5. Current chronic diarrhoea
6. Contraindication for corticosteroid administration
7. History of prior serious allergic or pseudo-allergic reaction
8. Any other serious illness or medical condition
9. Symptomatic peripheral neuropathy ≥ grade 2
10. Received mangafodipir ≤ 5 weeks before planned start of chemotherapy
11. Received any of the FOLFOX drugs ≤ 5 weeks before planned start of chemotherapy
12. Any plans of administered other anti-cancer therapy (including radiotherapy) concurrent with this study
13. Fertile females
14. Males with reproductive potential not implementing adequate contraception measures
15. Phaeochromocytoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Neutropenia | Before and after completion of one, two and/or three FOLFOX6-cycles

SECONDARY OUTCOMES:
Quality of Life | Before and after completion of one, two and/or three FOLFOX6-cycles

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Falkmer, MD, PhD, Principal Investigator — Länssjukhuset Ryhov
Locations (1):
- Onkologkliniken, Länssjukhuset Ryhov, Jönköping, Sweden

REFERENCES:
- [Background] Alexandre J, Nicco C, Chereau C, Laurent A, Weill B, Goldwasser F, Batteux F. Improvement of the therapeutic index of anticancer drugs by the superoxide dismutase mimic mangafodipir. J Natl Cancer Inst. 2006 Feb 15;98(4):236-44. doi: 10.1093/jnci/djj049. PMID 16478742
- [Background] Asplund A, Grant D, Karlsson JO. Mangafodipir (MnDPDP)-and MnCl2-induced endothelium-dependent relaxation in bovine mesenteric arteries. J Pharmacol Exp Ther. 1994 Nov;271(2):609-14. PMID 7965775
- [Background] Brurok H, Ardenkjaer-Larsen JH, Hansson G, Skarra S, Berg K, Karlsson JO, Laursen I, Jynge P. Manganese dipyridoxyl diphosphate: MRI contrast agent with antioxidative and cardioprotective properties? Biochem Biophys Res Commun. 1999 Jan 27;254(3):768-72. doi: 10.1006/bbrc.1998.0131. PMID 9920816
- [Background] Doroshow JH. Redox modulation of chemotherapy-induced tumor cell killing and normal tissue toxicity. J Natl Cancer Inst. 2006 Feb 15;98(4):223-5. doi: 10.1093/jnci/djj065. No abstract available. PMID 16478735
- [Background] Karlsson JO, Brurok H, Eriksen M, Towart R, Toft KG, Moen O, Engebretsen B, Jynge P, Refsum H. Cardioprotective effects of the MR contrast agent MnDPDP and its metabolite MnPLED upon reperfusion of the ischemic porcine myocardium. Acta Radiol. 2001 Nov;42(6):540-7. doi: 10.1080/028418501127347340. PMID 11736698
- [Background] Karlsson JO, Brurok H, Towart R, Jynge P. The magnetic resonance imaging contrast agent mangafodipir exerts antitumor activity via a previously described superoxide dismutase mimetic activity. Cancer Res. 2006 Jan 1;66(1):598; author reply 598. doi: 10.1158/0008-5472.CAN-05-2053. No abstract available. PMID 16397277